CLINICAL TRIAL: NCT03826615
Title: The Effect of Gabapentin Pretreatment on Hyperalgesia in Elderly Patients Undergoing Staged Bilateral Cataract Operations
Brief Title: Gabapentin Pretreatment for Staged Bilateral Cataract Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHSeo_gabapentin
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Hyperalgesia; Cataract Bilateral Nos
MeSH Terms: conditions — Hyperalgesia; Cataract | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin premedication group
  Interventions: Drug: Gabapentin
- No medication (No Intervention): Control group

INTERVENTIONS:
Drug: Gabapentin — Patients receive gabapentin 100mg orally for 3 times a day during the period of first and second cataract operations
  Arms: Gabapentin

SUMMARY:
To evaluate the effect of oral gabapentin premedication on hyperalgesia in elderly patients undergoing staged bilateral cataract operations under monitored anesthesia care

DETAILED DESCRIPTION:
It has been reported that patients with bilateral cataract complained more pain and discomfort during the second consecutive eye surgery compared to the first eye surgery.

Gabapentin is an anticonvulsant drug, which has been extended the use to perioperative analgesia, and anxiolysis.

Therefore, the investigators conducted this randomized, controlled study to evaluate the effects of gabapentin premedication on patients' subjective sensations, including intraoperative anxiety, perceptions of pain, and light sensitivity, in the second cataract operations.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 60 years, who undergoing staged bilateral cataract operations under monitored anesthesia care
* ASA physical status of I, II, and III

Exclusion Criteria:

* undergoing other eye operations together besides cataract operation
* patients with creatinin clearance lower than 30ml/min
* patients with CNS inhibitors medication
* patients with previous gabapentin medication
* pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Pain perception | during the operation
  intraoperative pain perception evaluated by VAS in first and second cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea